CLINICAL TRIAL: NCT04368793
Title: Intelligence-based Remote Pulmonary Rehabilitation and Efficacy Among Discharged COVID-19 Patients
Brief Title: Clinical Effects of Internet Assisted Pulmonary Rehabilitation of COVID-2019 Pneumonia Patients After Discharge
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: China-Japan Friendship Hospital (Other)
Collaborators: Wuhan lung Hospital (Unknown); Wuhan Central Hospital (Other); Wuhan University (Other); Ai You Foundation (Unknown)
Responsible Party: Principal Investigator, Hongtao Niu, Doctor, China-Japan Friendship Hospital
Other Study IDs: 2020-22-K17
Record Dates: First submitted 2020-04-23; First posted 2020-04-30 (Actual); Last update posted 2020-07-17 (Actual); Status verified 2020-07

CONDITIONS: COVID-2019 Pneumonia; Pulmonary Rehabilitation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Discharged COVID-19 patient cohort: All enrolled participants will be given 8 weeks (online 2 weeks + offline 6 weeks) pulmonary rehabilitation intervention, and will be followed up for at least one year, to assess their adherence and efficacy of the rehabilitation program.
  Interventions: Behavioral: Remote pulmonary rehabilitation

INTERVENTIONS:
Behavioral: Remote pulmonary rehabilitation — The pulmonary rehabilitation intervention includes respiratory exercise, barehanded aerobic training, exercise prescription of elastic band impedance training, respiratory muscle strength training, etc.

SUMMARY:
The noval coronavirus disease 2019 (COVID-19) would cause physical and psychological dysfunctions in infected patients. We expect that an intelligence-based remote pulmonary rehabilitation scheme could improve patients' health status after hospital discharge. The intelligence-based remote pulmonary rehabilitation program is designed in a real-world and prospective manner, aiming to evaluate the efficacy of rehabilitation among 200 patients in the epicenter of China (Wuhan City) according to their varied adherence. An eight-week rehabilitation scheme, including two weeks for physicians and physiotherapists remotely guided training, and six weeks for patient self-management, will be addressed. The primary outcome of current study is six-minute walking distance and lung function, and secondly respiratory muscle strength, physical fitness assessment, symptoms and quality of life, etc. will also be assessed. Recruited patients will be followed up at week 2, 4, 8 after enrollment and at month 1, 3, 6, 12 after the rehabilitation training completed, respectively. The study has been approved by the ethics committee of China-Japan Friendship Hospital and three participating centers in Wuhan City.

ELIGIBILITY:
Inclusion criteria:

* patients diagnosed as COVID-19 pneumonia according to the Chinese diagnostic criteria (Trial 7th Edition), aged 20 years or above;
* patients who did not participate in any other rehabilitation training scheme;
* patients who did not participate in any other intervention clinical trials;
* patients who signed the informed consent and were able to adhere to a long-term follow-up for at least one year.

Exclusion criteria:

* pregnant women;
* patients with previous mental disorders or undergoing mental health treatment;
* patients with previous personality disorder, intelligence disorder, brain injury or brain disease;
* patients with serious cardiovascular, cerebrovascular, neuromuscular and other systemic diseases or other diseases affecting physical activity;
* patients with tumors and underwent treatment.

One will be considered as withdrawal if consent is revoked, lost to follow-up, or unable to take the pulmonary rehabilitation scheme due to severe exacerbation, comorbidities, injury or trauma, etc.

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All discharged COVID-19 pneumonia patients who have signed the informed consent and met above eligibility criteria will be enrolled in this study.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2020-04-06 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Six-minute walking distance (6MWD) | One year
  Walking distance within six minutes
Pulmonary function | One year
  Forced expiratory volume in one second (FEV1), forced vital capacity (FVC), etc.

SECONDARY OUTCOMES:
Respiratory muscle strength | One year
  Maximal inspiratory pressure, maximal expiratory pressure, etc.
Physical fitness assessment | One year
  Two-minute walking test, short physical performance battery, grip strength of both upper limbs, knee extension strength of both lower limbs, etc.
Symptom | One year
  Modified British Medical Research Council (mMRC) dyspnea scale, etc.
Psychological evaluation | One year
  Self-training depression scale (SDS) and self-rating anxiety scale (SAS)
Quality of life | One year
  36-item short-form health survey (SF-36), etc.
Physical activity | One year
  International physical activity questionnaire (IPAQ)
Proportion of returning to society | One year
  Proportions of returning to routine work and normal life

CONTACTS AND LOCATIONS:
Overall Officials: Ting Yang, Prof., Principal Investigator — China-Japan Friendship Hospital
Locations (3):
- China (3):
  - Wuhan Lung Hospital, Wuhan, Hubei
  - Wuhan Central Hospital, Wuhan, Hubei
  - Zhongnan Hospital of Wuhan University, Wuhan, Hubei

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lei J, Yang L, Wen G, Qumu S, Ren X, Yang T. Pulmonary telerehabilitation and efficacy among discharged COVID-19 patients: Rational and design of a prospective real-world study. Clin Respir J. 2021 Nov;15(11):1158-1167. doi: 10.1111/crj.13422. Epub 2021 Aug 6. PMID 34260823